CLINICAL TRIAL: NCT03275688
Title: NanoSpectrometer Biomarker Discovery and Confirmation Study
Status: Terminated | Type: Observational
Why Stopped: Interim analysis showed sample size sufficient for final analysis
Sponsor: Johns Hopkins University (Other)
Collaborators: Nanobeak Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00121967
Record Dates: First submitted 2017-09-01; First posted 2017-09-07 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Lung Cancer
Keywords: lung cancer; volatile organic compound; screening; VOC; clinical trial
MeSH Terms: conditions — Lung Neoplasms | interventions — Breath Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breath sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stage 1 Lung Cancer (Case): These are the participants with identified stage 1 lung cancer.
  Interventions: Diagnostic Test: Breath Analysis
- Type 1 Control: These are participants who have similar clinical characteristics as our cases, but do not have any history of cancer.
  Interventions: Diagnostic Test: Breath Analysis
- Type 2 Control: These are housemates of the participants with stage 1 lung cancer (cases).
  Interventions: Diagnostic Test: Breath Analysis

INTERVENTIONS:
Diagnostic Test: Breath Analysis — Breath will be analyzed in all three groups using gas chromatography mass spectrometry.
  Other Names: Gas Chromatography Mass Spectrometry

SUMMARY:
This study will evaluate exhaled volatile organic compounds (VOC's) in the breath of participants with stage 1 lung cancer, their house-mates, and matched controls. The goal of the study is to identify VOC fingerprints that are only detectable in those with stage 1 lung cancer.

DETAILED DESCRIPTION:
Lung cancer is by far the leading cause of cancer death in the United States. More people die annually of lung cancer than of colon, breast, and prostate cancers combined. Worldwide it is already the leading cause of cancer death among males, and with smoking rates substantially higher in developing countries relative to the United States the worldwide burden of lung cancer is projected to increase considerably in the future.

For lung cancer, as for many cancers, early diagnosis allowing for full resection offers the greatest chance for long-term survival, but unfortunately these individuals currently constitute only a minority of the lung-cancer population. Screening technologies that allow for the earliest detection of lung cancer would therefore have tremendous potential to substantially improve outcomes. Recently, and for the first time, a screening test for lung cancer of high risk individuals has been recommended by the US Preventive Services Task Force, as well as others, for the reduction of lung cancer mortality. This recommendation was based primarily on the results of the National Lung Screening Trial (NLST) that randomized over 53,000 individuals considered at high risk for lung cancer to 3 annual screenings with either low-dose CT (LDCT) or a chest x-ray and then followed for a median of 6.5 years. In this study LDCT scanning was associated with a statistically significant 20% relative decrease in lung cancer mortality, and a smaller, but still significant 6.7% decrease in overall mortality. Despite these encouraging results of LDCT, as a screening tool it has substantial limitations. Beyond the costs, inconvenience and radiation exposure associated with LDCT, its performance characteristics are far from optimal. For example, nearly a quarter of the LDCT population had a positive screening test, with the vast majority - 96.4% - proving to be false-positive. With a positive predictive value of <4% LDCT screening will lead to a great number of unnecessary diagnostic procedures as well as substantial anxiety in the screened population and their family.

Breath analytics is a new and very promising tool for diagnosing lung cancer, as well as multiple other conditions. Previous studies identified that dog's heightened olfactory senses were able to detect cancer in an individual's breath with an accuracy of nearly 100%. Since then attempts have been made to mimic canine capabilities with "electronic noses" to detect and quantitate the nearly 3000 compounds, many in the parts per billion or even parts per trillion ranges, in exhaled breath. Early studies of these technologies support great potential as a diagnostic and screening tool. As a screening tool it could be ideal as it is noninvasive, painless and free of any undesirable side effects. In addition, new advances in nanotechnology have allowed these extremely sensitive detection technologies to be miniaturized to the point that they can be linked to a smartphone, providing future possibilities to almost continuously surveil individuals for the development of lung cancer and other life-threatening conditions. This study is concerned with comparing the concentrations of volatile organic compounds (VOCs) in the breath of lung cancer patients (cases) and lung-cancer-free individuals (controls).

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and over with diagnosed Stage 1 Lung Cancer (cases)
* Adults age 18 and over without Lung cancer (type 1 controls)
* Adults age 18 and over who live in the same environment as the cases (type 2 controls)

Exclusion Criteria N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of three groups. Our cases will be those who have been diagnosed with stage 1 lung cancer. Our type 1 controls will consist of participants who do not have lung cancer, but otherwise have similar clinical characteristics of our cases. the type 2 controls will be people who live in the same house as our stage 1 lung cancer patients (cases).
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2020-07-06 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Volatile organic compounds present in our cases but not controls. | 1.5 years
  Volatile organic compounds will be measured between the cases and both types of controls. We will report the different volatile organic compound fingerprints that are present in cases and not in controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lonny Yarmus, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No